CLINICAL TRIAL: NCT03512964
Title: A Pilot Study of Rapid HIV Treatment Initiation, Access and Engagement in Care (RHAE)
Brief Title: Rapid HIV Treatment Initiation, Access and Engagement in Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00110075; P30AI094189 (NIH)
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Results first posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-09

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — dolutegravir; Emtricitabine; tenofovir alafenamide; emtricitabine tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rapid HIV Treatment Initiation (Other): Initiation and reinitiation of antiretroviral therapy with dolutegravir 50 mg by mouth once daily and descovy 1 tablet by mouth once daily the same-day as HIV diagnosis and/or first clinic visit for people newly diagnosed with HIV and patients previously diagnosed with HIV but not on medications and not in care for over six months.
  Interventions: Drug: Dolutegravir 50 MG; Drug: Emtricitabine/Tenofovir Alafenamide 200 MG-25 MG Oral Tablet [DESCOVY]

INTERVENTIONS:
Drug: Dolutegravir 50 MG — Patients newly diagnosed with HIV or previously diagnosed with HIV and not on treatment or in care for at least six months will be given antiretroviral therapy starter packs containing dolutegravir (tivicay) 50 mg 1 tablet by mouth daily. Number of doses dispensed will be determined by the prescribing provider. Pill boxes will be given with each starter pack. At each clinic, patients are provided with 24/7 clinic contact information should he/she experience adverse side effects to medication and/or experience a medical emergency.
  Other Names: Tivicay
Drug: Emtricitabine/Tenofovir Alafenamide 200 MG-25 MG Oral Tablet [DESCOVY] — Patients newly diagnosed with HIV or previously diagnosed with HIV and not on treatment or in care for at least six months will be given antiretroviral therapy starter packs containing emtricitabine 200 mg/tenofovir alafenamide 25 mg (descovy) 1 tablet by mouth daily. Number of doses dispensed will be determined by the prescribing provider. Pill boxes will be given with each starter pack. At each clinic, patients are provided with 24/7 clinic contact information should he/she experience adverse side effects to medication and/or experience a medical emergency.
  Other Names: Descovy

SUMMARY:
The investigators propose to evaluate Rapid HIV Treatment Initiation in Baltimore in newly and previously diagnosed HIV-positive patients not in care through identification of barriers, facilitators and acceptability of Rapid HIV Treatment Initiation among newly and previously diagnosed HIV-positive patients not in care identified at the Johns Hopkins East Baltimore campus and at the Baltimore City Health Department sexually transmitted disease clinics. Using this data, a protocol for Rapid HIV Treatment Initiation among newly and previously diagnosed HIV-positive patients not in care identified at the Johns Hopkins East Baltimore campus and the Baltimore City Health Department sexually transmitted disease clinics will be developed and pilot tested. This pilot data will be used to design a multi-site study evaluating the effectiveness of Rapid HIV Treatment Initiation versus facilitated linkage to care. A model for Rapid HIV Treatment Initiation in Baltimore could be generalized to cities where the HIV epidemic has a similar demographic and risk profile such as Washington DC, Atlanta, and New York City.

DETAILED DESCRIPTION:
Prompt initiation of antiretroviral therapy to achieve and sustain viral suppression decreases the morbidity and mortality of HIV and greatly reduces the risk of transmission yet gaps in the care cascade persist. At current testing and treatment rates, an estimated 524,000 new infections and 375,000 deaths will occur between 2015 and 2025 in the US. Rates of HIV are unacceptably high among African Americans and men who have sex with men and a majority of new transmissions originate from patients previously diagnosed but not in care. To curb rates of infection and improve HIV-related outcomes, cities such as Baltimore, where the HIV epidemic predominately affects African Americans and men who have sex with men, must implement more effective ways to identify and treat all individuals with HIV. Compressing the treatment timeline by starting antiretroviral therapy at the time of diagnosis is known as rapid HIV treatment initiation. Early studies of Rapid HIV Treatment Initiation in newly diagnosed patients in South Africa and San Francisco showed significant improvement in care linkage, antiretroviral therapy initiation and time to viral suppression. Investigators propose to evaluate Rapid HIV Treatment Initiation in Baltimore in newly and previously diagnosed HIV-positive patients not in care through identification of barriers, facilitators and acceptability of Rapid HIV Treatment Initiation and pilot testing a protocol for Rapid HIV Treatment Initiation among newly and previously diagnosed HIV-positive patients not in care identified at the Johns Hopkins East Baltimore campus and at the Baltimore City Health Department sexually transmitted disease clinics. This pilot data will be used to design a multi-site study evaluating the effectiveness of Rapid HIV Treatment Initiation versus facilitated linkage to care. A model for Rapid HIV Treatment Initiation in Baltimore could be generalized to cities where the HIV epidemic has a similar demographic and risk profile such as Washington DC, Atlanta, and New York City.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 to 65 years of age
* English speaking
* Patients identified in the Hopkins Emergency Department, Hopkins John G. Bartlett Specialty Practice clinic or Baltimore City Health Department sexually transmitted disease clinics who are newly diagnosed with HIV (test positive by 3rd or 4th generation HIV test or detectable HIV viral load with no previously documented positive HIV test by medical record and/or self-report) and patients with previous HIV diagnosis but by self-report are not in care and not on antiretroviral therapy (> six months without HIV care or antiretroviral therapy)

Exclusion Criteria:

* Women who are currently pregnant or planning on becoming pregnant
* Adults lacking the capacity to consent
* Patients referred to HIV care outside of Johns Hopkins and/or Baltimore City Health Department Sexually Transmitted Diseases (STD) clinics
* Patients with estimated creatinine clearance <30 mL/min at last documented laboratory testing in the available medical record at site of referral, self-report of chronic kidney disease without documented creatinine within the last three months
* Patients who have pre-study documented HIV resistance mutations to dolutegravir or tenofovir alafenamide in the available medical record at site of referral or who self-report history of HIV resistance mutations. and susceptibility to dolutegravir and tenofovir alafenamide cannot be confirmed
* Patients with a contraindication to dolutegravir, tenofovir alafenamide and/or emtricitabine
* Patients on or in anticipation of starting a rifamycin medication (rifampin, rifabutin, or rifapentine) and/or carbamazepine
* Patients judged by clinic or study staff to be physically or emotionally unable to provide consent or participate in all study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2020-09-13 (Actual); Study Completion 2020-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Jones, MD, Principal Investigator — JohnsHopkins U
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Rapid HIV Treatment Initiation: Initiation and reinitiation of antiretroviral therapy with dolutegravir 50 mg by mouth once daily and descovy 1 tablet by mouth once daily the same-day as HIV diagnosis and/or first clinic visit for people newly diagnosed with HIV and patients previously diagnosed with HIV but not on medications and not in care for over six months.
  dolutegravir and descovy: Patients newly diagnosed with HIV or previously diagnosed with HIV and not on treatment or in care for at least six months will be given antiretroviral therapy starter packs containing dolutegravir (tivicay) 50 mg 1 tablet by mouth daily and emtricitabine 200 mg/tenofovir alafenamide 25 mg (descovy). Number of doses dispensed will be determined by the prescribing provider. Pill boxes will be given with each starter pack. At each clinic, patients are provided with 24/7 clinic contact information should he/she experience adverse side effects to medication and/or experience a medical emergency.
Period: Overall Study
Arm/Group | Rapid HIV Treatment Initiation
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rapid HIV Treatment Initiation
Number analyzed (Participants) | 32
Age, Continuous [Mean (Full Range); unit: years] | 40 [19 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1
  Black/African American | 30
  Native American | 1
  Alaskan Native | 0
  Pacific Islander | 0
  Other Asian | 0
  Some other race | 0
  Refused | 0
  Don't know | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Receive Rapid HIV Treatment Initiation
Description: Number of patients who do start Anti-retroviral Therapy (ART) the same day it is offered.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rapid HIV Treatment Initiation
Number analyzed (Participants) | 32
Participants | 32

2. Secondary Outcome: Rapid HIV Treatment Initiation Acceptability as Assessed by the Number of Patients Who Respond Yes to Starting ART Same Day
Description: Number of patients who respond yes to starting ART same day versus those who respond no in the survey.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Rapid HIV Treatment Initiation: Initiation and reinitiation of antiretroviral therapy with dolutegravir 50 mg by mouth once daily and descovy 1 tablet by mouth once daily the same-day as HIV diagnosis and/or first clinic visit for people newly diagnosed with HIV and patients previously diagnosed with HIV but not on medications and not in care for over six months.
  Rapid HIV treatment initiation and reinitiation: Patients newly diagnosed with HIV or previously diagnosed with HIV and not on treatment or in care for at least six months will be given antiretroviral therapy starter packs containing dolutegravir (tivicay) 50 mg 1 tablet by mouth daily and emtricitabine 200 mg/tenofovir alafenamide 25 mg (descovy) 1 tablet by mouth daily. Number of doses dispensed will be determined by the prescribing provider. Pill boxes will be given with each starter pack. At each clinic, patients are provided with 24/7 clinic contact information should he/she experience adverse side effects to medication and/or experience a medical emergency.
Arm/Group | Rapid HIV Treatment Initiation
Number analyzed (Participants) | 32
Participants | 32

3. Secondary Outcome: Number of Patients Offered Rapid HIV Treatment Initiation
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rapid HIV Treatment Initiation
Number analyzed (Participants) | 32
Participants | 32

4. Secondary Outcome: Number of Patients Who Accepted Rapid HIV Treatment Initiation
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rapid HIV Treatment Initiation
Number analyzed (Participants) | 32
Participants | 32

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Rapid HIV Treatment Initiation
All-Cause Mortality (participants affected / at risk) | 1/32
Serious Adverse Events (participants affected / at risk) | 1/32
Other Adverse Events (participants affected / at risk) | 1/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rapid HIV Treatment Initiation (N=32)
Death (Cardiac disorders) | 1 (1) — Participant fell down stairs and was found unresponsive. Upon Emergency Medical Service (EMS) arrival, patient was in cardiac arrest, asystole and resuscitation was unsuccessful. Event was more likely than not unrelated to research procedures.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rapid HIV Treatment Initiation (N=32)
Unnecessary ART initiation (Product Issues) | 1 (1) — HIV positive test at enrollment was false positive. Participant was exposed to antiretroviral therapy for 11 days despite not having HIV infection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT03512964/Prot_000.pdf